CLINICAL TRIAL: NCT03627299
Title: An Open-label Pilot Study to Determine the Safety and Efficacy of Fixed-dose Glecaprevir and Pibrentasvir Treatment in Hepatitis C Uninfected Recipients of Renal Transplants From Hepatitis C Infected Deceased Donors
Brief Title: Renal Transplants in Hepatitis C Negative Recipients With Nucleic Acid Positive Donors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00174409
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Results first posted 2020-08-24 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: End Stage Renal Disease; Hepatitis C
MeSH Terms: conditions — Kidney Failure, Chronic; Hepatitis C | interventions — glecaprevir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Deceased donor HCV RNA PCR+ (Experimental): Participants who receive a kidney from HCV RNA PCR + deceased donor will receive 300 mg glecaprevir/pibrentasivir 120 mg once daily by mouth for 4 weeks
  Interventions: Drug: 300mg glecaprevir/pibrentasivir 120mg

INTERVENTIONS:
Drug: 300mg glecaprevir/pibrentasivir 120mg — 300mg glecaprevir/pibrentasivir 120mg 4 weeks post-transplant
  Other Names: Mavyret

SUMMARY:
In this study, individuals without hepatitis C infection who are on the kidney transplant waitlist will receive a kidney from a deceased donor with hepatitis C infection and will be treated for hepatitis C at the same time. Treatment will include glecaprevir 300 mg / pibrentasvir 120 mg (G-P) administered on-call to the operating room for the renal transplant procedure and continued for 4 weeks post-renal transplant.

DETAILED DESCRIPTION:
In this study, individuals without hepatitis C infection who are on the kidney transplant waitlist will receive a kidney from a deceased donor with hepatitis C infection and will be treated for hepatitis C at the same time. Treatment will include glecaprevir 300 mg / pibrentasvir 120 mg (G-P) administered on-call to the operating room for the renal transplant procedure and continued for 4 weeks post-renal transplant. The participant will continue to be tested for Hepatitis C for 12 weeks post-treatment.

The primary hypothesis is that prophylactic treatment with glecaprevir/pibrentasvir before and after transplant will prevent the establishment of HCV infection in the recipients of kidneys from HCV-infected deceased donors. Based on the success of preliminary studies, the objective of the study is to evaluate the safety and efficacy of 4 weeks of G-P as prophylaxis for HCV D+/R- kidney transplant.

ELIGIBILITY:
Recipient Inclusion Criteria

* Participants ≥ 40 years old
* On the deceased donor kidney waitlist at Johns Hopkins Hospital
* Awaiting a first or second kidney transplant
* No available living kidney donors
* On hemodialysis or peritoneal dialysis or stage 5 chronic kidney disease defined as a glomerular filtration rate <15 ml/min for ≥ past 90 days
* HCV-uninfected (by both antibody and RNA PCR) and without any behavioral risk factors for contracting HCV other than being on hemodialysis
* Calculated panel reactive anti-human leukocyte antigen antibody (cPRA) below 80%

Recipient Exclusion Criteria

* Plan to receive a multi-organ transplant
* Plan to receive a dual kidney transplant (including en bloc)
* Prior solid organ transplant
* Participating in another study that involves an intervention or investigational product
* Plan to receive a blood type incompatible kidney
* History of human immunodeficiency (HIV), hepatitis C (HCV), or active hepatitis B (HBV) infection, defined as being on active antiviral treatment for HBV, detectable hepatitis B surface Ag or detectable hepatitis B DNA
* Unable to safely substitute or discontinue a medication that is contraindicated with the study medication
* Psychiatric or physical illness that in the opinion of the investigator would make it unsafe to proceed with transplantation or interfere with the ability of the subject to participate in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Durand, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Peer reviewed publications

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 11 participants who signed consent, 10 received organ offers from HCV+ deceased donors. The remaining participant did not receive an offer before enrollment in the study closed.
Period: Overall Study
Arm/Group | Deceased Donor HCV RNA PCR+
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 67 [40 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Primary Cause of Renal Failure [Count of Participants; unit: Participants]
  Hypertension | 4
  Polycystic Kidney Disease | 2
  Glomerulonephritis | 2
  Nephrolithiasis | 1
  Reflux Nephropathy | 1
Blood Type [Count of Participants; unit: Participants]
  O | 4
  A or AB | 5
  B | 1

OUTCOME MEASURES:

1. Primary Outcome: Viral Response at Week 12
Description: This is the number of participants with undetectable hepatitis C RNA in the blood at 12 weeks after stopping treatment. Proportion of kidney transplant recipients with HCV RNA < Lower Limit Of Quantification (LLOQ) at week 12
Time Frame: 12 weeks after completing therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Number of Participants With Grade 3 or Higher Treatment-related Adverse Events Related to the Use of G-P
Description: Proportion of participants with grade 3 or higher treatment-related adverse events (AE) as assessed by US Department of Health and Human Services Common Terminology of AEs version 4. An AE is an unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5. Grade 3 Severe or medically significant but not life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE. The investigator will determine if the AE is related to the treatment.
Time Frame: 4 weeks after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Participants | 0

3. Secondary Outcome: Viral Response at 1 Week
Description: This is the number of participants with undetectable hepatitis C RNA in the blood at 1 week after stopping treatment. Proportion of kidney transplant recipients with HCV RNA < Lower Limit Of Quantification (LLOQ) at week 1
Time Frame: 1 week after completing therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Participants | 8

4. Secondary Outcome: Viral Response at 2 Weeks
Description: This is the number of participants with undetectable hepatitis C RNA in the blood at 2 weeks after stopping treatment. Proportion of kidney transplant recipients with HCV RNA < Lower Limit Of Quantification (LLOQ) at week 2
Time Frame: 2 weeks after completing therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Participants | 10

5. Secondary Outcome: Viral Response at 4 Weeks
Description: This is the number of participants with undetectable hepatitis C RNA in the blood at 4 weeks after stopping treatment. Proportion of kidney transplant recipients with HCV RNA < Lower Limit Of Quantification (LLOQ) at week 4
Time Frame: 4 weeks after completing therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Participants | 10

6. Secondary Outcome: Viral Response at 8 Weeks
Description: This is the number of participants with undetectable hepatitis C RNA in the blood at 8 weeks after stopping treatment. Proportion of kidney transplant recipients with HCV RNA < Lower Limit Of Quantification (LLOQ) at week 8
Time Frame: 8 weeks after completing therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Participants | 10

7. Secondary Outcome: Antibody Development
Description: Number of kidney transplant recipients that become reactive for HCV antibody
Time Frame: week 12 after discontinuation of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Participants | 9

8. Secondary Outcome: T-cell Response at Baseline
Description: Measurement of t-cell response to HCV peptides, a marker of acute hepatitis C infection. This categorizes participants into no T-cell response, T-cell response to 1 peptide, T-cell response to 2 peptides and T-cell response to 3 peptides.
Time Frame: Baseline prior to induction therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Participants
  No T-cell response at baseline | 6
  T-cell response to 1 peptide at baseline | 1
  T-cell response to 2 peptides at baseline | 2
  T-cell response to 3 peptides at baseline | 1

9. Secondary Outcome: T-cell Response at 12 Weeks
Description: as for outcome 8
Time Frame: Week12 after discontinuation of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Participants
  No T-cell response at 12 weeks | 5
  T-cell response to 1 peptide at 12 weeks | 3
  T-cell response to 2 peptides at 12 weeks | 1
  T-cell response to 3 peptides at 12 weeks | 1

10. Secondary Outcome: Kidney Function at 6 Months
Description: Serum creatinine mg/dL at 6 months following transplantation
Time Frame: 6 months following transplant
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
mg/dL | 1.32 [0.8 to 2.0]

11. Secondary Outcome: Kidney Function at 12 Months
Description: Serum creatinine mg/dL at 12 months following transplantation
Time Frame: 12 months following transplant
Population: One participant did not have serum creatinine checked at 12 months post-transplantation.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 9
mg/dL | 1.33 [0.79 to 4.12]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 12 months from initiation of treatment
Arm/Group | Deceased Donor HCV RNA PCR+
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deceased Donor HCV RNA PCR+ (N=10)
Renal Vein Thrombosis (Renal and urinary disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Perinephric Fluid Collection (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT03627299/Prot_SAP_000.pdf